CLINICAL TRIAL: NCT02116374
Title: Correlation Between Microbiota Biodiversity of HIV Seropositive Patients With Their Clinical and Immunological Status (ANRS EP 55 MICROGUT).
Brief Title: Physiopathology Study of the Microbiota Biodiversity of HIV Seropositive Patients
Acronym: MICROGUT
Status: Completed | Type: Observational
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS EP55 MICROGUT; 2014-A00216-41 (Other: ANSM)
Record Dates: First submitted 2014-04-15; First posted 2014-04-16 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: HIV-1 Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool sample
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- HIV-1 patients
  Interventions: Other: Physiopathology study

INTERVENTIONS:
Other: Physiopathology study

SUMMARY:
The bacterial diversity of HIV patients digestive microbiota seropositive is poorly understood, it remains to be defined.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 or more.
* Patients with a confirmed diagnosis of HIV infection 1.
* Patient who signed an informed consent form.
* Patient affiliated or beneficiary of a social security system.

Exclusion Criteria:

* Patient known to be suffering from inflammatory bowel disease (Crohn's disease or ulcerative colitis).
* Patient HIV-2 or HIV-1/HIV-2 co-infected
* Patient having received immunotherapy
* Patient participating in another research.
* Pregnant women, parturient or lactating person under guardianship, or deprived of liberty by a judicial or administrative decision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-1 seropositive patients
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2014-12; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Proportion and type of OTU (Operational Taxonomic Unit) assigned to the rank of phylum genus and species of bacteria in the intestinal microbiota of HIV-1 seropositive patients. | Baseline

SECONDARY OUTCOMES:
Proportion and OTU types in the gastrointestinal microbiota of HIV-1 seropositive patients compared to the general population | Baseline
Proportion and OTU types in the gastrointestinal microbiota of HIV-1 seropositive patients based on CD4, viral load, the Elite controller status, antiretroviral and antibiotic treatment and the existence of invasive bacterial infections. | Baseline
Proportion and OTU types in the gastrointestinal microbiota of HIV-1 seropositive patients based on inflammation parameters (IL-6, TNF-a, IP-10), CRPus, CD14 and integrity of the epithelial barrier (I-FABP). | Baseline
Transcriptomic analysis in the groups that present differences in the microbiota and analysis of lymphocyte populations Th17 and Treg. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Didier Raoult, MD, Principal Investigator — IHU Méditerranée infection
Locations (4):
- France (4):
  - Centre Henri Mondor, Créteil
  - Service de Médecine Interne et Immunologie Clinique, Le Kremlin-Bicêtre
  - IHU Méditerranée Infection; Hôpital Nord, AP-HM, Marseille
  - Service de maladies Infectieuses, Marseille